CLINICAL TRIAL: NCT02440620
Title: Cardiac Toxicity in Medical Treatment of Breast Cancer
Acronym: CaTOB
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ann Banke, MD, Ph.d.-student, Odense University Hospital
Other Study IDs: S-20140090
Record Dates: First submitted 2015-04-29; First posted 2015-05-12 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure; Breast Cancer
Keywords: Heart failure related to medical treatment of breast cancer
MeSH Terms: conditions — Heart Failure; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be analyzed for N-terminal proBNP and ultra-sensitive TnT. Targeted sequencing of a limited number of well-known genes related to heart failure will be conducted and analysis of potential future biomarkers related to heart failure is possible from blood samples stored in a biobank.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will describe the epidemiology including prognosis of heart failure related to treatment with anthracycline and trastuzumab for breast cancer.

In a prospective study Human Epidermal Growth Factor Receptor 2 (HER2) positive breast cancer patients scheduled for trastuzumab treatment at Odense University Hospital, will be offered advanced echocardiographic examination, test of bio-markers and genetic markers for the purpose of investigating if early identification of patients in particular risk of developing heart failure is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HER2 positive breast cancer
* Adjuvant treatment with trastuzumab

Exclusion Criteria:

* Left ventricle ejection fraction (LVEF) <50%
* Chronic or persistent atrial fibrillation
* History of moderate or severe valvular heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2 positive breast cancer in adjuvant treatment with trastuzumab.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Global longitudinal strain by two dimentional speckle tracking. | Change in outcome from initiation of trastuzumab treatment and after 3,6, and 9 month.
Ratio between the mitral E velocity and early diastolic maximum global strain rate (E/SRE). | Change in outcome from initiation of trastuzumab treatment and after 3,6, and 9 month.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Moeller, MD, DMsc, Study Director — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Denmark